CLINICAL TRIAL: NCT01633359
Title: The Randomly Controlled Clinical Trial of the Association Between Very Small Embryonic-like Stem Cells and the Prognosis of Coronary Artery Disease Patients
Brief Title: The Association Between Very Small Embryonic-like Stem Cells and the Prognosis of Coronary Artery Disease Patients
Acronym: VSEL-CAD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ji Huang (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor-Investigator, Ji Huang, Attending Physician of Cardiology, Beijing Anzhen Hospital
Organization: Beijing Anzhen Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRAVEL-CAD
Record Dates: First submitted 2012-05-31; First posted 2012-07-04 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive statin (Experimental): 1. Fifty CAD subjects will receive intensive Atorvastatin administration and 50 CAD patients receiving the routine Atorvastatin administration as controls.
  2. All subjects will receive the follow-up for 1 year, and peripheral blood VSELs, SDF-1/CXCR4 are tested, and the MACE (major adverse cardiovascular events) are recorded including angina, repeat myocardial infarction, repeat revascularization, major organ dysfunction, and death.
  3. the Intensive Atorvastatin protocol indicates that 80mg Atorvastatin will be administrated before CAG, and then are followed with 20mg Atorvastatin during the entire study period.
  Interventions: Drug: Intensive statin
- Routine statin (Experimental): 1. Fifty CAD subjects will receive intensive Atorvastatin administration and 50 CAD patients receiving the routine Atorvastatin administration as controls.
  2. All subjects will receive the follow-up for 1 year, and peripheral blood VSELs, SDF-1/CXCR4 are tested, and the MACE (major adverse cardiovascular events) are recorded including angina, repeat myocardial infarction, repeat revascularization, major organ dysfunction, and death.
  3. the Routine Atorvastatin protocol indicates that 20mg Atorvastatin daily during the entire study period.
  Interventions: Drug: Routine statin

INTERVENTIONS:
Drug: Intensive statin — the Intensive Atorvastatin protocol indicates that once 80mg Atorvastatin will be administrated before CAG, and then will be followed with 20mg Atorvastatin daily during the entire study period.
  Other Names: Intensive Atorvastatin
  Arms: Intensive statin
Drug: Routine statin — the Routine Atorvastatin protocol indicates that 20mg Atorvastatin daily during the entire study period.
  Other Names: Routine Atorvastatin.
  Arms: Routine statin

SUMMARY:
Hypothesis: Peripheral blood Very Small Embryonic-like Stem Cells (VSELs) are different in coronary artery disease (CAD) patients from those without CAD, which might account for the benefits of Atorvastatin in CAD patients.

DETAILED DESCRIPTION:
1. Hypothesis: The VSELs might be mobilized in the situation of cardiac ischemia in CAD patients. In addition, the benefits derived from Atorvastatin administration in CAD patients may be related to VSELs via sCD40L-SDF1/CXCR4 signal pathway.
2. The number and function of peripheral blood VSELs in CAD patients compared with the controls.

   1. Included patients: including 200 CAD patients receiving coronary angiography (CAG) as positive subjects, 100 as control who are negative for CAG.
   2. The IRB approve and all subjects sign the informed consent.
   3. All subjects will receive the detection and analysis of the peripheral blood VSELs, including VSEL number, immigration capability after sCD40L administration.
   4. All subjects will receive the follow-up for 1 year, and the MACE (major adverse cardiovascular events) are recorded including angina, repeat myocardial infarction, repeat revascularization, major organ dysfunction, and death.
   5. the association between VSELs and MACE in CAD patients will be statistically analyzed.
3. Atorvastatin administration improves the prognosis of CAD patients through exerting impacts on VSELs

   1. Included patients: including 200 CAD patients receiving coronary angiography as positive subjects, 100 as control who are negative for coronary angiography.
   2. The IRB approve and all subjects sign the informed consent.
   3. Fifty CAD subjects will receive intensive Atorvastatin administration and 50 CAD patients receiving the routine Atorvastatin administration as controls.
   4. All subject will receive the follow-up for 1 year, and peripheral blood VSELs, SDF-1/CXCR4 are tested, and the MACE (major adverse cardiovascular events) are recorded including angina, repeat myocardial infarction, repeat revascularization, major organ dysfunction, and death.
   5. the Intensive Atorvastatin protocol indicates that 80mg Atorvastatin will be administrated before CAG, and then are followed with 20mg Atorvastatin during the entire study period.
   6. the Routine Atorvastatin protocol indicates that 20mg Atorvastatin daily during the entire study period.

ELIGIBILITY:
Inclusion Criteria:

* CAD patients receiving coronary angiography (CAG) as positive subjects, 100 as control who are negative for CAG.

Exclusion Criteria:

* Infectious diseases, immunologically mediated disease, serious liver diseases, serious kidney diseases, malignant tumor, thrombocytopenia, pregnancy, occluded peripheral arterial diseases, bleeding or blood transfusion in the latest 2 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-07; Primary Completion 2012-12 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Number of peripheral blood VSELs | during 1 year after enrollment
  All subject will receive the follow-up for 1 year, and peripheral blood VSELs are counted.

SECONDARY OUTCOMES:
MACE | During 1 year in the study period
  All subject will receive the follow-up for 1 year, and the MACE (major adverse cardiovascular events) are recorded including angina, repeat myocardial infarction, repeat revascularization, major organ dysfunction, and death.

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Yan Qian, MD,PhD, Study Director — Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Wojakowski W, Tendera M, Kucia M, Zuba-Surma E, Paczkowska E, Ciosek J, Halasa M, Krol M, Kazmierski M, Buszman P, Ochala A, Ratajczak J, Machalinski B, Ratajczak MZ. Mobilization of bone marrow-derived Oct-4+ SSEA-4+ very small embryonic-like stem cells in patients with acute myocardial infarction. J Am Coll Cardiol. 2009 Jan 6;53(1):1-9. doi: 10.1016/j.jacc.2008.09.029. PMID 19118716